CLINICAL TRIAL: NCT07098273
Title: Restoring Manual Dexterity in Multiple Sclerosis: A Feasibility Study Combining Muscle Electrostimulation and Transcranial Magnetic Stimulation To Enhance Neuroplasticity
Brief Title: Improving Hand Movement and Coordination in People With Multiple Sclerosis Using Transcranial Magnetic Stimulation (TMS) and Muscle Electrostimulation (FES) To Support Manual Dexterity and Daily Function
Acronym: MANTRAStim
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MANTRAStim-SC; 2024/R-Multi/010 (Other Grant/Funding Number: Fondazione Italiana Sclerosi Multipla)
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Hand Dexterity; Technology-based Rehabilitation; Functional Electrical Stimulation; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Pilot, controlled, multicenter, national, non-profit experimental study with parallel arms, double-blind (evaluator and participant), without the use of drugs or medical devices.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS-FES group (Experimental): Before movement execution, the hand area of the primary motor cortex will be stimulated using active repetitive TMS (rTMS). Subsequently, FES will be applied to assist the subject's voluntary movements during task-oriented therapy.
  Interventions: Device: TMS and FES- based rehabilitation
- FES group (Active Comparator): Before movement execution, the hand area of the primary motor cortex will be stimulated using sham TMS. Subsequently, FES will be applied to assist the subject's voluntary movements during task-oriented therapy.
  Interventions: Device: FES-based rehabilitation

INTERVENTIONS:
Device: TMS and FES- based rehabilitation — Each subject will receive 15 individual sessions (45 minutes each, 3 times per week for 5 weeks) of task-based hand and arm exercises.
  Before movement execution, the hand area of the primary motor cortex will be stimulated using active rTMS. The rTMS protocol will use intermittent theta burst stimulation (iTBS), which delivers bursts of 3 pulses at 50 Hz every 200 ms (5 Hz) for 2 seconds, followed by 8 seconds of rest, totaling 600 pulses in ~3 minutes. The hand area will be identified as the optimal site for eliciting a motor evoked potential (MEP) in the abductor digiti minimi (ADM) muscle, contralateral to the dominant limb, with the lowest possible stimulation intensity.
  Subsequently, FES will be applied to assist the subject's voluntary movements during the task-oriented activities. The stimulation will be triggered based on the achievement of the electromyographic (EMG) threshold of the selected muscles.
  Arms: TMS-FES group
Device: FES-based rehabilitation — Each subject will receive 15 individual sessions (45 minutes each, 3 times per week for 5 weeks) of task-based hand and arm exercises.
  Before movement execution, the TMS coil will be positioned over the hand areas of the primary motor cortex, but tilted away from the scalp so as to produce a sound similar to the real intervention, but at a low intensity, without inducing current in the cortex.
  FES will then be applied to assist the patient's voluntary movements during the task-oriented activities. The stimulation will be triggered based on the achievement of the electromyographic (EMG) threshold of the selected muscles.
  Arms: FES group

SUMMARY:
The goal of this interventional study is to test whether combining transcranial magnetic stimulation (TMS) with functional electrical stimulation (FES) can improve hand and upper limb function in adults with Multiple Sclerosis (MS).

The clinical trial aims to determine the following points:

1. Whether TMS combined with FES produces greater effects compared to FES alone.
2. Changes in brain and muscle activity related to hand function after treatment.
3. Specific clinical or neurophysiological factors that predict who will benefit most from the intervention. Researchers will compare the TMS-FES group (receiving brain magnetic stimulation and muscle electrostimulation) with the FES group (receiving only muscle electrostimulation) to assess whether TMS provides additional benefits in improving upper limb function

Participants will:

* Be assigned to a group (TMS-FES group or FES group)
* Attend 15 sessions (45 minutes each, 3 times per week for 5 weeks) of task-based hand and arm exercises, during which FES, or TMS and FES, will be administered to the participant.
* Undergo assessments before, after, and 3 months after training to measure hand function, brain and muscle responses, fatigue, and daily activity performance.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic disease of the central nervous system associated with various neurological deficits, including motor impairments that negatively affect autonomy and quality of life. Among these, a significant symptom is reduced manual dexterity, which affects approximately 75% of patients and can interfere with activities of daily living (ADLs), leading to job loss and the need for assistance. This deficit, considered an indicator of disability in progressive MS, stems from altered sensorimotor integration and damage to various neural structures.

In recent years, non-invasive brain stimulation techniques, particularly Transcranial Magnetic Stimulation (TMS), have shown potential in measuring changes in cortical excitability and improving MS symptoms. TMS is a sensitive method for detecting cortical alterations and assessing corticospinal tract function through motor evoked potentials (MEPs), which are reliable biomarkers of disease progression. Moreover, studies and meta-analyses suggest that repetitive TMS (rTMS) may have therapeutic effects on cognitive deficits, spasticity, and fatigue in MS patients. In particular, stimulation of the primary motor cortex (M1) through rTMS has been shown to improve hand movement speed, although the effect dissipates quickly-typically after about 20 minutes.

To prolong these benefits, integrating TMS with Functional Electrical Stimulation (FES) could be an effective strategy. FES stimulates muscles through external surface electrical impulses to counteract the contractile inefficiency typical of MS and may further enhance residual motor function during voluntary exercises by promoting adaptive neuroplasticity. FES is already widely used in gait rehabilitation for MS, with positive effects on muscle strength and quality of life.

However, the application of FES for hand rehabilitation remains less explored, despite recommendations in favor of its investigation.

There is an urgent therapeutic need for non-pharmacological approaches to address upper limb and hand deficits, given their disabling impact on the MS population. Recent guidelines suggest exploring FES as an adjunct to traditional rehabilitation therapy to enhance its effects and improve access to rehabilitation for patients with muscle weakness.

The investigators hypothesize that the combination of TMS and FES may increase cortical excitability, reduce fatigue, and improve motor learning, leading to more effective recovery. The proposed study will assess the feasibility of a rehabilitation protocol based on these technologies, analyzing their effects on manual dexterity and on the central and peripheral neurophysiological correlates of motor recovery.

Furthermore, the investigators aim to identify predictive biomarkers of functional recovery, with the goal of personalizing rehabilitation pathways and optimizing therapeutic interventions for MS.

In this study, 30 individuals with MS are planned to be recruited, divided into the TMS-FES experimental group and the FES group. In the TMS-FES group, the primary motor cortex hand areas will be stimulated with active repetitive TMS before motor execution, while the FES group will receive sham TMS stimulation. Both groups will receive muscular electrical stimulation to assist voluntary movements during task-oriented activities.

The training will consist of three sessions per week, each lasting 45 minutes, for a total of 15 sessions. The investigators will measure variables such as age, gender, clinical status, fatigue, health perception, TMS-based biomarkers, and upper limb muscle synergies in all participants before and after the training. The investigators will investigate long-term effects on motor control, kinematic movement, and daily functional mobility three months after the end of the training through instrumental assessments and self-administered questionnaire.

20 healthy subjects are planned to be recruited, who will serve as the normative reference for the instrumental analysis assessments. The subjects will take part in a single data collection session, during which upper limb kinematics and EMG signals will be recorded while performing instrumented tasks from the Action Research Arm Test (ARAT) used for instrumental evaluation.

ELIGIBILITY:
Inclusion Criteria:

* age >18;
* diagnosis of MS (according to McDonald criteria);
* stable disease course without a worsening greater than 1 point on the Expanded Disability Status Scale (EDSS) in the past 4 months;
* right-handed;
* score on the Box and Block test lower than the normative value adjusted for sex and age +2 standard deviations;
* score on the cerebellar functional system of the EDSS scale <2;
* ability to provide written informed consent.

Exclusion Criteria:

* score on the Mini-Mental State Examination <24;
* Beck Depression Inventory-II >19;
* other neurological or orthopedic conditions that would interfere with upper limb exercises;
* contraindications to the application of TMS: history of epilepsy or non-febrile seizures; presence of metallic or electronic implants in the cranial or cervical region; presence of pacemakers or implantable defibrillators; severe uncontrolled psychiatric disorders (e.g., psychosis, mania); current or suspected pregnancy;
* contraindications to the application of FES: skin integrity issues at the site of electrode placement; implanted electronic devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
9-Hole Peg Test (9HPT) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  The 9-Hole Peg Test evaluates manual dexterity and fine motor function of the upper limb. The test consists in taking pegs from a container, one by one, and place them into the holes on the board, as quickly as possible, using only the hand being evaluated. Pegs then have to be removed from the holes, one by one, and be placed back into the container.
  Score is given according to the number of seconds it takes for the patient to complete the test or alternatively, the number of pegs placed in 50 or 100 seconds.

SECONDARY OUTCOMES:
Box and Block Test (BBT) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. The BBT goal is to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds. The score is determined by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period. Higher scores on the test indicate better gross manual dexterity
Arm Function in Multiple Sclerosis Questionnaire (AMSQ) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  The Arm Function in Multiple Sclerosis Questionnaire (AMSQ) is a unidimensional 31-item questionnaire for measuring arm function in Multiple Sclerosis. Each item asks about the extent to which MS has limited the individual's ability to perform specific daily activities in the past two weeks and is rated on a scale, from 1 (not at all) to 6 (unable to perform this activity). The total score is calculated by summing the scores for all items, and higher scores indicate greater limitations.
Symbol Digit Modalities Test (SDMT) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  The Symbol Digit Modalities Test (SDMT) examines processing speed and sustained attention by primarily assessing complex visual scanning and tracking. Using a reference key, the test taker has 90 seconds to pair specific numbers with given geometric figures. Responses can be written or given orally, and administration time is just five minutes for either response mode.
12-Item Short Form Survey (SF-12) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  The 12-Item Short Form Survey (SF-12) is a self-reported outcome measure assessing the impact of health on an individual's everyday life. Patients fill out a 12-question survey covering physical and mental health domain, which is then scored by a clinician or researcher. The responses are scored using a standardized algorithm to calculate two summary scores: the Physical Component Summary (PCS-12) and the Mental Component Summary (MCS-12). These scores are interpreted using a norm-based scoring system, with a mean of 50 and a standard deviation of 10 in the general population. Higher scores generally indicate better health.
Fatigue Scale of Motor and Cognitive Functions (FSMC) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  The Fatigue Scale of Motor and Cognitive Functions (FSMC) is a 20-item scale developed as a measure of cognitive and motor fatigue for people with MS. The responses to the items are summed to create separate scores for motor and cognitive fatigue, as well as a total fatigue score. Higher scores generally indicate greater fatigue.
Intrinsic Motivation Inventory (IMI) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  The Intrinsic Motivation Inventory (IMI) is a multidimensional measurement device intended to assess participants' subjective experience related to a target activity in laboratory experiments. The instrument yields six subscale scores assessing participants': interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice while performing a given activity.
System Usability Scale (SUS) | After (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks).
  The System Usability Scale (SUS) is a well-established and reliable tool for assessing the usability of rehabilitation technologies. It consists of 10 statements that evaluate aspects such as ease of use, intuitiveness, and effectiveness. Participants rate each statement on a 5-point scale, ranging from "strongly disagree" to "strongly agree." The responses are then calculated to produce a final usability score out of 100.

OTHER OUTCOMES:
Surface Electromyography (EMGs) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  Surface Electromyography (EMGs) is a non-invasive tool able to assess muscular electrical activity during the execution of active movements using electrodes applied on the skin surface. Muscular contraction amplitude will be recorded from 24 sensors placed on upper limbs (12 sensors/limb), during the execution of motor acts. Then, the difference between patient's and observed model's temporal dynamic of muscular contraction will be chosen as EMG outcome.
Body Kinematics | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  Kinematics of the upper limb and trunk will be recorded using a 9-camera optoelectronic system during 3D motor acts. The system will measure the 3D coordinates of spherical markers attached to body landmarks to compute trunk, shoulder, elbow, wrist, and finger angles. Data processing will provide measures of deviations from physiological movement.
Motor Evoked Potential (MEP) | Before (T0) and after (T1) the rehabilitation treatment (15 sessions of 45 minutes each, 3 times per week for 5 weeks), and at 3 months from T1 (T2).
  In order to detect changes in corticospinal function and neural plasticity induced by the intervention, the neurophysiological protocol consists of recording motor evoked potentials (MEPs) from the abductor digiti minimi (ADM) muscle of the upper limb, using a focused coil with neuronavigated positioning on the scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Lencioni, PhD, Principal Investigator — IRCCS "Santa Maria Nascente" - Fondazione Don Gnocchi
Locations (2):
- Italy (2):
  - Fondazione Italiana Sclerosi Multipla, Genova, Italy
  - IRCCS "Santa Maria Nascente" - Fondazione Don Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Shared data will comprise only IPD used in results publication. Data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication with no end date
Access Criteria: Request should be addressed to the principal investigator or the corresponding author of the publication.

REFERENCES:
- [Background] Sirbu CA, Thompson DC, Plesa FC, Vasile TM, Jianu DC, Mitrica M, Anghel D, Stefani C. Neurorehabilitation in Multiple Sclerosis-A Review of Present Approaches and Future Considerations. J Clin Med. 2022 Nov 27;11(23):7003. doi: 10.3390/jcm11237003. PMID 36498578
- [Background] Severijns D, Lamers I, Kerkhofs L, Feys P. Hand grip fatigability in persons with multiple sclerosis according to hand dominance and disease progression. J Rehabil Med. 2015 Feb;47(2):154-60. doi: 10.2340/16501977-1897. PMID 25268997
- [Background] Sampson P, Freeman C, Coote S, Demain S, Feys P, Meadmore K, Hughes AM. Using Functional Electrical Stimulation Mediated by Iterative Learning Control and Robotics to Improve Arm Movement for People With Multiple Sclerosis. IEEE Trans Neural Syst Rehabil Eng. 2016 Feb;24(2):235-48. doi: 10.1109/TNSRE.2015.2413906. Epub 2015 Mar 24. PMID 25823038
- [Background] Reeves BC, Wells GA, Waddington H. Quasi-experimental study designs series-paper 5: a checklist for classifying studies evaluating the effects on health interventions-a taxonomy without labels. J Clin Epidemiol. 2017 Sep;89:30-42. doi: 10.1016/j.jclinepi.2017.02.016. Epub 2017 Mar 27. PMID 28351692
- [Background] Neira VE, Niemietz TD, Farrell JW 3rd. THE EFFECTS OF EXERCISE TRAINING ON UPPER EXTREMITY FUNCTION FOR PERSONS WITH MULTIPLE SCLEROSIS: A SYSTEMATIC REVIEW. J Rehabil Med Clin Commun. 2022 Sep 29;5:2306. doi: 10.2340/jrmcc.v5.2306. eCollection 2022. PMID 36249930
- [Background] Lo DF, Palhang M, Gawash A, Zia H, Goodwin BJ, Patel K, White CP. Unlocking Therapeutic Potential: The Role of Theta Burst Stimulation in Multiple Sclerosis Management. Prim Care Companion CNS Disord. 2024 Apr 18;26(2):23r03645. doi: 10.4088/PCC.23r03645. PMID 38684013
- [Background] Leodori G, Mancuso M, Maccarrone D, Tartaglia M, Ianniello A, Certo F, Baione V, Ferrazzano G, Malimpensa L, Belvisi D, Pozzilli C, Berardelli A, Conte A. Neural bases of motor fatigue in multiple sclerosis: A multimodal approach using neuromuscular assessment and TMS-EEG. Neurobiol Dis. 2023 May;180:106073. doi: 10.1016/j.nbd.2023.106073. Epub 2023 Mar 9. PMID 36906073
- [Background] Koch G, Rossi S, Prosperetti C, Codeca C, Monteleone F, Petrosini L, Bernardi G, Centonze D. Improvement of hand dexterity following motor cortex rTMS in multiple sclerosis patients with cerebellar impairment. Mult Scler. 2008 Aug;14(7):995-8. doi: 10.1177/1352458508088710. Epub 2008 Jun 23. PMID 18573820
- [Background] Kim Y, Steiner P. Quasi-Experimental Designs for Causal Inference. Educ Psychol. 2016;51(3-4):395-405. doi: 10.1080/00461520.2016.1207177. Epub 2016 Sep 2. PMID 30100637
- [Background] Kamm CP, Uitdehaag BM, Polman CH. Multiple sclerosis: current knowledge and future outlook. Eur Neurol. 2014;72(3-4):132-41. doi: 10.1159/000360528. Epub 2014 Jul 30. PMID 25095894
- [Background] Jonsdottir J, Perini G, Ascolese A, Bowman T, Montesano A, Lawo M, Bertoni R. Unilateral arm rehabilitation for persons with multiple sclerosis using serious games in a virtual reality approach: Bilateral treatment effect? Mult Scler Relat Disord. 2019 Oct;35:76-82. doi: 10.1016/j.msard.2019.07.010. Epub 2019 Jul 20. PMID 31352180
- [Background] Jones S, Man WD, Gao W, Higginson IJ, Wilcock A, Maddocks M. Neuromuscular electrical stimulation for muscle weakness in adults with advanced disease. Cochrane Database Syst Rev. 2016 Oct 17;10(10):CD009419. doi: 10.1002/14651858.CD009419.pub3. PMID 27748503
- [Background] Huertas-Hoyas E, Maximo-Bocanegra N, Diaz-Toro C, Montes-Diez R, Perez-Corrales J, Sanchez-Herrera-Baeza P, Martinez-Piedrola RM, Garcia-Bravo C, Sanchez-Camarero C, Perez-de-Heredia-Torres M. A Descriptive Cross-Sectional Study of Manipulative Dexterity on Different Subtypes of Multiple Sclerosis. Occup Ther Int. 2020 Apr 28;2020:6193938. doi: 10.1155/2020/6193938. eCollection 2020. PMID 32425718
- [Background] Fan J, Fu H, Xie X, Zhong D, Li Y, Liu X, Zhang H, Zhang J, Huang J, Li J, Jin R, Zheng Z. The effectiveness and safety of repetitive transcranial magnetic stimulation on spasticity after upper motor neuron injury: A systematic review and meta-analysis. Front Neural Circuits. 2022 Nov 8;16:973561. doi: 10.3389/fncir.2022.973561. eCollection 2022. PMID 36426136
- [Background] Conradsson D, Ytterberg C, von Koch L, Johansson S. Changes in disability in people with multiple sclerosis: a 10-year prospective study. J Neurol. 2018 Jan;265(1):119-126. doi: 10.1007/s00415-017-8676-8. Epub 2017 Nov 20. PMID 29159465
- [Background] Chruzander C, Johansson S, Gottberg K, Einarsson U, Fredrikson S, Holmqvist LW, Ytterberg C. A 10-year follow-up of a population-based study of people with multiple sclerosis in Stockholm, Sweden: changes in disability and the value of different factors in predicting disability and mortality. J Neurol Sci. 2013 Sep 15;332(1-2):121-7. doi: 10.1016/j.jns.2013.07.003. Epub 2013 Jul 26. PMID 23896259
- [Background] Bashir S, Mizrahi I, Weaver K, Fregni F, Pascual-Leone A. Assessment and modulation of neural plasticity in rehabilitation with transcranial magnetic stimulation. PM R. 2010 Dec;2(12 Suppl 2):S253-68. doi: 10.1016/j.pmrj.2010.10.015. PMID 21172687
- [Background] Barnighausen T, Tugwell P, Rottingen JA, Shemilt I, Rockers P, Geldsetzer P, Lavis J, Grimshaw J, Daniels K, Brown A, Bor J, Tanner J, Rashidian A, Barreto M, Vollmer S, Atun R. Quasi-experimental study designs series-paper 4: uses and value. J Clin Epidemiol. 2017 Sep;89:21-29. doi: 10.1016/j.jclinepi.2017.03.012. Epub 2017 Mar 30. PMID 28365303
- [Background] Ayache SS, Riachi N, Ahdab R, Chalah MA. Effects of Transcranial Direct Current Stimulation on Hand Dexterity in Multiple Sclerosis: A Design for a Randomized Controlled Trial. Brain Sci. 2020 Mar 23;10(3):185. doi: 10.3390/brainsci10030185. PMID 32210025
- [Background] Alenazy M, Daneshgar Asl S, Petrigna L, Feka K, Alvarez E, Almuklass AM, Enoka RM. Treatment with electrical stimulation of sensory nerves improves motor function and disability status in persons with multiple sclerosis: A pilot study. J Electromyogr Kinesiol. 2021 Dec;61:102607. doi: 10.1016/j.jelekin.2021.102607. Epub 2021 Oct 13. PMID 34710779